CLINICAL TRIAL: NCT03771482
Title: Education of Providers on Prescribing Best Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Matthew McEvoy, Professor of Anesthesiology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 190371
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid module first then fluid (Active Comparator): The providers in this arm will first receive daily information and questions related to opioid use for eight weeks and then daily information and questions related to intravenous fluid prescribing for five weeks.
  Interventions: Behavioral: Quiztime modules
- Fluid module first then opioid (Active Comparator): The providers in this arm will first receive daily information and questions related to intravenous fluid prescribing for five weeks and then daily information and questions related to opioid use for eight weeks.
  Interventions: Behavioral: Quiztime modules

INTERVENTIONS:
Behavioral: Quiztime modules — Text Messaging or Email system

SUMMARY:
This study aims to evaluate the impact of spaced education, delivered via a smartphone application, on provider prescribing patterns.

DETAILED DESCRIPTION:
As part of a medical center educational initiative at Vanderbilt University Medical Center (VUMC), two educational modules will be sent to prescribing providers through either email or short message service (SMS) text messaging. The first educational module consists of a set of multiple choice questions concerning best practices for prescribing intravenous fluids in the inpatient and perioperative setting. This module is based upon recent literature and specifically derived from the results of the Isotonic Solutions and Major Adverse Renal Events Trial (SMART) and Saline Against Lactated Ringer's or Plasma-Lyte in the Emergency Department (SALT-ED) trial, both published in the New England Journal of Medicine in 2018 and led by Vanderbilt investigators. Similarly, a second educational module concerning evidence-based pain management and opioid prescribing practices will be distributed via email or SMS text messaging.

Participants will receive one question per day. If the participant does not answer the question correctly, they will receive the opportunity to attempt the question again after reviewing evidence-based education. All questions have been curated and reviewed by a panel of experts and piloted within VUMC for feasibility and acceptability. Key concepts are repeated in each module and questions are strategically ordered throughout each module to accomplish spaced education.

ELIGIBILITY:
Inclusion Criteria:

* All inpatient prescribing providers

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Median morphine milligram equivalents (MME) per opioid prescription | 8 months
  By extracting prescribing data for opioids from the electronic health records
Percentage of orders for balanced intravenous (IV) fluid solutions (i.e. not normal saline) | 8 months
  By extracting prescribing data for intravenous fluids from the electronic health records

SECONDARY OUTCOMES:
Chloride levels in patients receiving intravenous fluid orders from a provider enrolled in the study | 8 months
  By extracting chloride level data from the electronic health records
Potassium levels in patients receiving intravenous fluid orders from a provider enrolled in the study | 8 months
  By extracting potassium level data from the electronic health records
Major Adverse Kidney Events by 30 days (MAKE 30) in patients receiving intravenous fluid orders from a provider enrolled in the study | 30 days
  By extracting data from the electronic health records
Length of stay for patients receiving an intravenous fluid order or an opioid prescription from a provider enrolled in the study. | 8 months
  By extracting length of stay data from the electronic health records
Length of stay in the intensive care unit (ICU) for patients receiving an intravenous fluid order or an opioid prescription from a provider enrolled in the study | 8 months
  By extracting ICU length of stay from the electronic health records
Median number of pills per prescription for patients receiving an opioid prescription from a provider enrolled in the study | 8 months
  By extracting medication data from the electronic health records
Percent of opioid prescriptions (inpatient) that also had a scheduled (not pro re nata (PRN)) non-opioid (APAP, nonsteroidal anti-inflammatory drugs (NSAIDs), gamma-Aminobutyric acid (GABA), muscle relaxant, etc.) | 8 months
  By extracting medication data from the electronic health records
Percent of opioid prescriptions (discharge) that also had a scheduled (not PRN) non-opioid (APAP, NSAIDs, GABA, muscle relaxant, etc.) | 8 months
  By extracting medication data from the electronic health records
Number of Rapid Response Team calls (RRT s) indexed to the number of patients cared for per prescriber (evaluated by level of engagement of the learner with QuizTime) | 8 months
  By extracting RRT calls from the electronic health records

CONTACTS AND LOCATIONS:
Overall Officials: Matthew McEvoy, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Data dictionaries and individual participant data that underlie the results reported after de-identification will be available.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 3 months after publication for 5 years
Access Criteria: Researchers who provide a methodologically sound proposal that has been approved by the Vanderbilt Institutional Review Board and the study executive committee.

REFERENCES:
- [Derived] McEvoy MD, Dear ML, Buie R, Edwards DA, Barrett TW, Allen B, Robertson AC, Fowler LC, Hennessy C, Miller BM, Garvey KV, Bland RP 3rd, Fleming GM, Moore D, Rice TW, Bernard GR, Lindsell CJ; Vanderbilt Learning Healthcare System Platform Investigators and the Vanderbilt Committee on Opioid Monitoring and Stewardship. Effect of Smartphone App-Based Education on Clinician Prescribing Habits in a Learning Health Care System: A Randomized Cluster Crossover Trial. JAMA Netw Open. 2022 Jul 1;5(7):e2223099. doi: 10.1001/jamanetworkopen.2022.23099. PMID 35881398
- [Derived] McEvoy MD, Dear ML, Buie R, Fowler LC, Miller B, Fleming GM, Moore D, Rice TW, Bernard GR, Lindsell CJ; Vanderbilt Learning Healthcare System Investigators. Embedding Learning in a Learning Health Care System to Improve Clinical Practice. Acad Med. 2021 Sep 1;96(9):1311-1314. doi: 10.1097/ACM.0000000000003969. PMID 33570841